CLINICAL TRIAL: NCT00400712
Title: Client Centred 'Tune-ups': do They Enhance Community Reintegration and Mobility in Stroke Survivors?
Brief Title: Client Centred 'Tune-ups': do They Enhance Community Reintegration After Stroke?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Dr. Brenda Brouwer, Principle investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS SRA 5974
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Stroke
Keywords: mobility; strength; balance; function; reintegration; community
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): natural progression post-stroke
- Intervention (Experimental): two weeks of goal directed intensive physical rehabilitation therapy at 6 months (and one year)
  Interventions: Behavioral: physical rehabilitation

INTERVENTIONS:
Behavioral: physical rehabilitation — two weeks intensive physical rehabilitation
  Arms: Intervention

SUMMARY:
Once discharged from hospital many stroke survivors deteriorate medically, physically and in their mobility function and many report their level of function and quality of life to be poor 12 months after inpatient rehabilitation. There is an identified need for follow-up examinations of community dwelling stroke survivors to monitor changes in function and it has been suggested that maintenance therapy could curtail declines in function. The purpose of this trial is to determine whether brief periods of intense client-centered rehabilitation therapy (tune-ups) provided at 6 month intervals can alter the natural progression of impairment (physical capacity), function and community reintegration following stroke.

DETAILED DESCRIPTION:
The extent to which impairment (physical capacity) and function influence community reintegration is unclear. One of the challenges is that physical parameters change over time as does the person's awareness and perception of what activities are important to be able to engage in at the community level. Interventions have led to gains in physical capacity, function and community reintegration, but the benefits have been shown to dissipate within three to six months. It has been suggested that maintenance therapy (tune-ups) for stroke survivors post-discharge could prevent or curtail decline in function of aging stroke survivors and enhance quality of life and well being; constructs that relate strongly to community reintegration. This study will determine whether tune-ups can alter the time course and magnitude of changes in physical capacity and function and their influence on community reintegration. Stroke survivors discharged from rehabilitation will be followed for a 15 month period with laboratory or home assessments conducted at 3 month intervals. Assessors will be blind to whether the subject is receiving a tune up. Evaluations conducted after the tune-up at 9 months and 12 months post-discharge will allow us to determine if the tune-up effectively reduced physical impairment, improved function and resulted in better community reintegration compared to control.

ELIGIBILITY:
Inclusion Criteria:

* first major unilateral hemispheric stroke,
* english speaking,
* adequate verbal communication,
* discharged home or residential care

Exclusion Criteria:

* serious comorbidities (eg. cancer, mobility limiting arthritis, leg amputation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-12; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda J Brouwer, PhD, Principal Investigator — Queen's University; Jayne Garland, Ph.D, Principal Investigator — Western University, Canada
Locations (2):
- Canada (2):
  - Queen's University School of Rehabilitation Therapy, Kingston, Ontario
  - School of Physical Therapy, University of Western Ontario, London, Ontario

REFERENCES:
- [Derived] Brouwer B, Bryant D, Garland SJ. Effectiveness of Client-Centered "Tune-Ups" on Community Reintegration, Mobility, and Quality of Life After Stroke: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Jul;99(7):1325-1332. doi: 10.1016/j.apmr.2017.12.034. Epub 2018 Apr 3. PMID 29412167
- [Derived] Cohen JW, Ivanova TD, Brouwer B, Miller KJ, Bryant D, Garland SJ. Do Performance Measures of Strength, Balance, and Mobility Predict Quality of Life and Community Reintegration After Stroke? Arch Phys Med Rehabil. 2018 Apr;99(4):713-719. doi: 10.1016/j.apmr.2017.12.007. Epub 2018 Jan 6. PMID 29317222

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: no intervention, natural history following stroke
- Intervention: two weeks of goal directed intensive physical rehabilitation therapy aimed at improving mobility at 6 months (and one year)
Period: Overall Study
Arm/Group | Control | Intervention
Started | 52 | 51
Completed | 35 | 35
Not Completed | 17 | 16
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 11 | 12
Not completed — Physician Decision | 5 | 4

BASELINE CHARACTERISTICS:
Population: Hemiparetic stroke (hemorrhagic or ischemic), first ever associated with residual deficits/impairments (i.e. full recovery from previous stoke if applicable)
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (1.8) | 62.7 (1.7) | 62.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 30 | 24 | 54
Admission Functional Independence [Mean (Standard Deviation); unit: units on a scale] — The Functional Independence Measure (FIM) is an instrument that provides an indication of an individual's level of disability and their ability to perform activities of daily living (ADL). Eighteen (18) ADL-related motor and cognitive items are each rated on an ordinal scale ranging from complete dependence (1) to complete independence (7). The total FIM score ranges from 18 (lowest) to 126 (highest, complete independence).
  units on a scale | 96.2 (23.4) | 100.5 (22.1) | 98.4 (22.7)
Balance ability [Mean (Standard Deviation); unit: units on a scale] — The Berg Balance Scale (BBS) is composed of 14 items that require the individual to perform specific balance tasks ranging from basic (e.g. sit-to-stand, unsupported standing) to more difficult (e.g. standing on one leg). Each item is scored on an ordinal scale from 0 (unable to perform) to 4 (able to complete independently and/or safely). The total score ranges from 0 (lowest) to 56 (highest).
  units on a scale | 45.4 (13.5) | 47.8 (11.9) | 46.6 (12.8)
living setting pre-stroke [Number; unit: participants]
  private home | 51 | 50 | 101
  other | 1 | 1 | 2
mental status (MMSE) [Mean (Standard Deviation); unit: points] — The Mini-Mental State Exam (MMSE) is a screening tool for cognitive impairment. It is an 11 item questionnaire that tests five areas of cognitive function including orientation, attention and recall. A maximum score is 30 (total number of correct responses, 1 to 5 per question). A score of 23 or lower indicates cognitive impairment.
  points | 28 (0) | 28 (0) | 28 (0)
paretic side [Number; unit: participants]
  left hemiparesis | 37 | 29 | 66
  right hemiparesis | 15 | 22 | 37

OUTCOME MEASURES:

1. Primary Outcome: Subjective Index of Physical and Social Outcome (SIPSO)
Description: The SIPSO is a 10-item measure developed specifically for stroke that includes a Physical Integration Subscale relating to activities and daily living and a Social Integration subscale relating to social adaptation. Each item is assessed on an ordinal scale from 0 (cannot perform the task or activity/completely dissatisfied) to 4 (no difficultly/completely satisfied) such that the minimum score is 0 and the maximum for each subscale is 20 and the maximum total score is 40 (sum of subscales). The total score reflects reintegration.
Time Frame: baseline and 1 year
Population: those who completed 1 year testing
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 35 | 35
scores on a scale
  baseline | 26.6 (1.1) | 26.8 (1.2)
  one year | 29.7 (0.8) | 30.1 (0.8)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.44, ANCOVA; Examined whether there were differences between groups at 1 year with baseline measures serving as the covariate with a two-sided alpha of 0.05

2. Secondary Outcome: Mobility Function
Description: Timed up and go - participants stand from a seated position on a chair with armrests, walk 3 meters, turn and return to a seated position (measured in seconds)
Time Frame: baseline and 1 year
Population: those still enrolled at primary endpoint (one year)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control | Intervention
Number analyzed (Participants) | 35 | 35
seconds
  Baseline | 23.1 (3.4) | 19.9 (3.4)
  One year | 18.7 (2.0) | 19.7 (2.0)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.83, ANCOVA — Examined whether there were differences between groups at 1 year with baseline measures serving as the covariate with a two-sided alpha of 0.05

3. Secondary Outcome: Physical Capacity
Description: 6 minute walk test (6MWT). Subjects were instructed to walk as far as possible over 6 minutes with rests as needed and the distance traveled was recorded.
Time Frame: baseline and 12 months
Population: all those enrolled at primary endpoint - 1 year
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Control | Intervention
Number analyzed (Participants) | 35 | 35
meters
  Baseline | 258.9 (23.9) | 285.1 (25.1)
  One year | 332.0 (19.2) | 338.1 (20.2)
Statistical Analysis 1: Comparison: Control vs Intervention; ANCOVA - comparing absolute measures and including baseline as co-variate; Test type: Superiority or Other; p = 0.45, ANCOVA

4. Secondary Outcome: Health-related Quality of Life - Physical
Description: The SF-36 contains 36 questions pertaining to 8 health-related domains (physical and social function, emotional and physical limitation (role-emotional/role-physical), mental health, vitality, bodily pain, and general health). The derivation of the Physical component summary (PCS) score takes into account the physical health domains (physical function, role-physical and bodily pain) and scores self-reported physical health on a scale from 0 to 100, where 0 is the lowest rating of physical health and 100, the highest or best.
Time Frame: baseline and one year
Population: those enrolled at primary endpoint (one year)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Control | Intervention
Number analyzed (Participants) | 35 | 35
points
  Baseline | 35.7 (1.2) | 36.4 (1.3)
  One year | 42.0 (1.1) | 40.3 (1.2)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.72, ANCOVA; adjusted for baseline values

5. Secondary Outcome: Health-related Quality of Life - Mental
Description: The SF-36 contains 36 questions pertaining to 8 health-related domains (physical and social function, emotional and physical limitation (role-emotional/role-physical), mental health, vitality, bodily pain, and general health). The derivation of the Mental component summary (MCS) score takes into account the mental health domains (social function, role-emotional and mental health) and scores self-reported mental health on a scale from 0 to 100, where 0 is the lowest rating of mental health and 100, the highest.
Time Frame: baseline and one year
Population: those enrolled at 1 year (primary endpoint)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Control | Intervention
Number analyzed (Participants) | 35 | 35
points
  Baseline | 48.0 (2.0) | 49.3 (1.6)
  One year | 52.8 (1.3) | 51.2 (1.4)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.60, ANCOVA; controlled for baseline values

6. Primary Outcome: Subjective Index of Social Integration (Subscale of SIPSO)
Description: see Subjective Index of Physical and Social Outcome (SIPSO) above
Time Frame: baseline and one year
Population: those who completed 1 year testing
Measure: Mean (Standard Deviation); unit: points on a scale
Groups:
- Control: no intervention, natural progression post-stroke
- Intervention: two weeks of goal directed intensive physical rehabilitation therapy aimed at improving mobility at 6 months .
Arm/Group | Control | Intervention
Number analyzed (Participants) | 35 | 35
points on a scale
  Baseline | 13.8 (0.6) | 14.0 (0.7)
  One year | 14.4 (0.5) | 14.7 (0.7)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.66, ANCOVA — [p-value comment as in outcome 2, analysis 1]

7. Primary Outcome: Subjective Index of Physical Integration (Subscale of SIPSO)
Description: see 'Subjective Index of Physical and Social Outcome (SIPSO) above
Time Frame: baseline and one year
Population: those who completed 1 year testing
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 35 | 35
points on a scale
  Baseline | 12.9 (0.7) | 12.8 (0.8)
  One year | 15.2 (0.4) | 15.4 (0.4)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.78, ANCOVA — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: over one year
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 0/52 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No